CLINICAL TRIAL: NCT05294003
Title: Prevalence of West Nile Virus and Usutu Virus Serum Antibodies in Dutch Bird Ringers
Brief Title: West Nile Virus Seroprevalence Under Bird Ringers
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); Leiden University (Other); Netherlands Institute of Ecology (Unknown)
Responsible Party: Principal Investigator, Chiara de Bellegarde, Principal Investigator, Leiden University Medical Center
Other Study IDs: P20.112
Record Dates: First submitted 2022-02-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: West Nile Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In August 2020, West Nile Virus (WNV) was isolated from a live common whitethroat for the first time in The Netherlands. Follow-up sampling showed that the virus could also be detected in mosquitos from the same location during at least a whole month of sampling. On 15 October 2020, one case of West Nile virus infection has been reported in a man who was likely infected in the Utrecht region. This is the first time that a locally acquired human case of WNV infection has been reported in The Netherlands. Six additional cases have been identified, one of which from the region Arnhem. West Nile virus infection is a mosquito-borne zoonosis. The disease, which has spread across the Northern Hemisphere in the past three decades, is now found on an annual basis in many European countries where the centre of gravity lies in Southern-European countries. Recently, WNV was reported for the first time in Germany. The virus is transmitted among birds through the bite of infected mosquitoes and incidentally infects humans and other mammals, such as horses. Around 80% of human WNV infections are asymptomatic. The most common clinical presentation is West Nile fever but, older people and immunocompromised persons are at higher risk of developing neuro-invasive disorders (West Nile neuroinvasive disease). Currently, there are no prophylaxis or specific treatment against the disease in humans. In addition, Usutu virus (USUV) was detected in The Netherlands in 2016. USUV is another flavivirus, related to WNV, and also capable of infecting humans. Disease associated with USUV infection in humans appears to be milder and only limited number of cases have been identified. During their bird catching activities, bird ringers are intensively exposed to mosquito bites at the natural habitat of the birds and at the same time of the day when mosquitoes are particularly active. The aim of this study is therefore to determine the prevalence of WNV and USUV serum antibodies in bird ringers in The Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Carrying-out bird ringing activities during spring, summer or early autumn 2020 in The Netherlands

Exclusion Criteria:

* Not willing to participate in this study
* Using medication interfering with antibodies production
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bird ringers from the Netherlands (about 580 licensed ringers and about 100 additional trainees or helpers)
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
The proportion of individuals with neutralising antibodies against WNV by region | One blood sample collected between June and September 2021
The proportion of individuals with neutralising antibodies against USUV by region | One blood sample collected between June and September 2021

SECONDARY OUTCOMES:
The proportion of individuals with IgM antibodies against WNV | One blood sample collected between June and September 2021
The proportion of individuals with IgG antibodies against WNV | One blood sample collected between June and September 2021
The proportion of individuals with IgM antibodies against USUV | One blood sample collected between June and September 2021
The proportion of individuals with IgG antibodies against USUV | One blood sample collected between June and September 2021

CONTACTS AND LOCATIONS:
Overall Officials: Chiara de Bellegarde, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Centre (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sikkema RS, Schrama M, van den Berg T, Morren J, Munger E, Krol L, van der Beek JG, Blom R, Chestakova I, van der Linden A, Boter M, van Mastrigt T, Molenkamp R, Koenraadt CJ, van den Brand JM, Oude Munnink BB, Koopmans MP, van der Jeugd H. Detection of West Nile virus in a common whitethroat (Curruca communis) and Culex mosquitoes in the Netherlands, 2020. Euro Surveill. 2020 Oct;25(40):2001704. doi: 10.2807/1560-7917.ES.2020.25.40.2001704. PMID 33034280
- [Background] Ziegler U, Santos PD, Groschup MH, Hattendorf C, Eiden M, Hoper D, Eisermann P, Keller M, Michel F, Klopfleisch R, Muller K, Werner D, Kampen H, Beer M, Frank C, Lachmann R, Tews BA, Wylezich C, Rinder M, Lachmann L, Grunewald T, Szentiks CA, Sieg M, Schmidt-Chanasit J, Cadar D, Luhken R. West Nile Virus Epidemic in Germany Triggered by Epizootic Emergence, 2019. Viruses. 2020 Apr 15;12(4):448. doi: 10.3390/v12040448. PMID 32326472
- [Background] Gaibani P, Rossini G. An overview of Usutu virus. Microbes Infect. 2017 Jul-Aug;19(7-8):382-387. doi: 10.1016/j.micinf.2017.05.003. Epub 2017 Jun 8. PMID 28602915
- [Background] Rijks JM, Kik ML, Slaterus R, Foppen R, Stroo A, IJzer J, Stahl J, Grone A, Koopmans M, van der Jeugd HP, Reusken C. Widespread Usutu virus outbreak in birds in the Netherlands, 2016. Euro Surveill. 2016 Nov 10;21(45):30391. doi: 10.2807/1560-7917.ES.2016.21.45.30391. PMID 27918257
- [Background] Oude Munnink BB, Munger E, Nieuwenhuijse DF, Kohl R, van der Linden A, Schapendonk CME, van der Jeugd H, Kik M, Rijks JM, Reusken CBEM, Koopmans M. Genomic monitoring to understand the emergence and spread of Usutu virus in the Netherlands, 2016-2018. Sci Rep. 2020 Feb 18;10(1):2798. doi: 10.1038/s41598-020-59692-y. PMID 32071379
- See also: Rijksinstituut voor Volksgezondheid en Milieu, Ministerie van Volksgezondheid, Welzijn en Sport. Eerste patiënt in Nederland met westnijlvirus — https://www.rivm.nl/nieuws/eerste-patient-in-nederland-met-westnijlvirus
- See also: European Center for Disease Prevention and Control. Factsheet about West Nile fever [Internet]. Stockholm: ECDC; 2020 — https://www.ecdc.europa.eu/en/west-nile-fever/facts/factsheet-about-west-nile-fever
- See also: Rijksinstituut voor Volksgezondheid en Milieu, Ministerie van Volksgezondheid, Welzijn en Sport. Westnijlkoorts — https://www.rivm.nl/westnijlkoorts